CLINICAL TRIAL: NCT07267702
Title: Cultural Adaptation of a One-Day Online Cognitive Behavioral Therapy Group Workshop for Postpartum Depression in Türkiye: A Pilot Randomized Controlled Trial
Brief Title: Postpartum 1-Day CBT Pilot Study (Türkiye)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Büşra Kalaça, Assistant Doctor, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 09.2025.118
Record Dates: First submitted 2025-11-14; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Postpartum Depression
Keywords: Cognitive Behavioral Therapy; Online Intervention; Cultural Adaptation; Women, Gender and Mental Health; Feasibility Study; Randomized Controlled Trial; Psychotherapy; Mood Disorders; Depressive Disorder; Behavioral Disciplines and Activities; Depression, Postpartum
MeSH Terms: conditions — Depression, Postpartum; Coitus; Psychological Well-Being; Mood Disorders; Depressive Disorder; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned (1:1) to one of two parallel groups: (1) an intervention group receiving the culturally adapted one-day online CBT-based workshop, or (2) a control-usual care group.
Masking Description: This is an open-label pilot randomized controlled trial. Participants and facilitators cannot be blinded due to the nature of the behavioral intervention. However, outcome assessors and data analysts will remain blinded to group assignment to reduce potential assessment and analysis bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-Day Online CBT-Based Workshop (Experimental): Participants in this arm will receive the culturally adapted one-day online CBT-based workshop within the first month after enrollment, in addition to standard postpartum care.
  Interventions: Behavioral: One-Day Online CBT-Based Workshop
- Control Usual Care (No Intervention): Participants assigned to the control arm will continue to receive standard postnatal care from their healthcare providers.

INTERVENTIONS:
Behavioral: One-Day Online CBT-Based Workshop — The online workshop is a culturally adapted, one-day group intervention designed for women experiencing postpartum depression in Türkiye. Adapted from a validated Canadian model, it is delivered online by trained facilitators and includes approximately six hours of instruction. The four-module program provides brief psychoeducation about postpartum depression, introduces core cognitive and behavioral skills (e.g., cognitive restructuring, problem-solving, behavioral activation, assertiveness), and concludes with goal setting and action planning. Teaching methods include short lectures, group discussions, and role-plays. Regular breaks are included, and each participant receives a Turkish-language booklet to support engagement.
  Arms: One-Day Online CBT-Based Workshop

SUMMARY:
This pilot randomized controlled trial aims to evaluate the feasibility, acceptability, and preliminary effects of a culturally adapted, one-day online Cognitive Behavioral Therapy (CBT)-based group workshop for women with postpartum depression in Türkiye. The intervention was adapted from a validated model developed in Ontario, Canada, using Bernal's cultural adaptation framework.

Participants will be randomly assigned in a 1:1 ratio to either a workshop group, who will receive the one-day online CBT-based workshop within the first month after enrollment, or a control group who will continue to receive usual postpartum care throughout the study period. Data will be collected at baseline and at the 3-month follow-up using the Edinburgh Postnatal Depression Scale (EPDS), Patient Health Questionnaire-9 (PHQ-9), Generalized Anxiety Disorder-7 (GAD-7), the Frequency of Actions and Thoughts Scale (FATS), and the TÜRBAD Satisfaction Questionnaire (TÜRBAD-SQ).

The study will assess feasibility indicators including recruitment, randomization procedures, completion of study questionnaires, retention through the 3-month follow-up, and adherence to the one-day workshop. Acceptability and preliminary changes in depressive, anxiety, and cognitive-behavioral outcomes will also be explored.

This pilot trial represents the first culturally adapted, one-day online CBT-based group intervention for postpartum depression in Türkiye and will inform the design of a future large-scale randomized controlled trial.

DETAILED DESCRIPTION:
Postpartum depression (PPD) is a major public health concern affecting approximately one in five women worldwide and nearly one in five mothers in Türkiye. Despite its high prevalence, access to brief, evidence-based, and scalable psychological interventions remains limited, particularly in low- and middle-income settings. Untreated PPD increases the risk of chronic depression, impaired mother-infant bonding, and adverse emotional, behavioral, and developmental outcomes in children.

Cognitive Behavioral Therapy (CBT) is recommended as a first-line treatment for mild to moderate depression in the perinatal period; however, conventional CBT typically requires 12-15 weekly sessions, which can be difficult for new mothers due to caregiving demands, time limitations, and social isolation. Group-based interventions promote normalization and peer support but remain relatively inaccessible. Therefore, brief, structured, and scalable models are urgently needed.

A one-day CBT-based group workshop developed in Ontario, Canada has demonstrated feasibility, acceptability, and effectiveness in reducing postpartum depression. This study represents one of the first efforts to culturally adapt and evaluate this workshop for women in Türkiye. The adaptation followed Bernal's cultural adaptation framework to ensure conceptual, linguistic, and contextual relevance. All intervention materials were refined and finalized for pilot implementation following this adaptation phase.

This pilot randomized controlled trial aims to evaluate the feasibility, acceptability, and preliminary effectiveness of the culturally adapted one-day online CBT-based workshop among women with postpartum depressive symptoms in Türkiye. Sixty participants aged 18-45 years within the first postpartum year and with an Edinburgh Postnatal Depression Scale (EPDS) score ≥10 will be randomly assigned (1:1) to one of two groups: (1) a workshop group, who will receive the one-day online CBT-based workshop within the first month after enrollment; or (2) a control group, who will continue to receive usual postpartum care.

Eligible participants will be women aged 18-45 years who are within one year postpartum, have an EPDS score ≥10, are literate in Turkish, and have access to a stable internet connection. Exclusion criteria include current psychotic, bipolar, organic mental, or substance use disorders; a severe depressive episode requiring immediate clinical intervention; active suicidal ideation or intent; serious medical or neurological conditions that impair participation; or having an infant with a life-threatening congenital condition.

Assessments will be administered at baseline and at three months and will include the EPDS, Patient Health Questionnaire-9 (PHQ-9), Generalized Anxiety Disorder-7 (GAD-7), Frequency of Actions and Thoughts Scale (FATS), and the TÜRBAD Satisfaction Questionnaire (TÜRBAD-SQ). Although some Turkish validation studies suggest an EPDS cut-off of 12-13, a threshold of 10 was selected to align with international postpartum mental health research and to capture clinically relevant depressive symptoms.

Participants will be recruited through Marmara University clinical settings and community outreach channels.

Data collection and randomization will be conducted using REDCap (Research Electronic Data Capture) to ensure secure data management and methodological rigor. Findings from this pilot study will inform refinement of the intervention procedures, feasibility targets, and outcome measures, and will guide the development of a future large-scale randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18-45 years
* Having an infant aged 1-12 months
* Presence of clinically relevant postpartum depressive symptoms (EPDS ≥10)
* Literate in Turkish (able to read and write)
* Access to a stable internet connection
* Willing and able to provide informed consent

Exclusion Criteria:

* Current psychotic, bipolar, organic mental, or substance use disorder
* Severe depressive episode or impaired judgment due to psychiatric illness
* Active suicidal ideation or intent
* Medical or neurological condition preventing participation (e.g., dementia, intellectual disability, severe hearing or visual impairment)
* Infant with a life-threatening congenital disorder

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Recruitment Feasibility (Number of Participants Enrolled) | 6 months
  The total number of participants successfully enrolled in the study will be recorded to assess recruitment feasibility. The target is to enroll 60 participants (30 intervention, 30 control) within six months.
Proportion of Participants Completing All Study Questionnaires (EPDS, PHQ-9, GAD-7, FATS, TSQ) | Baseline and 3 months
  This outcome will assess the proportion of participants who complete all required study questionnaires (EPDS, PHQ-9, GAD-7, FATS, and TÜRBAD-SQ) at both baseline and the 3-month follow-up. Completion will be calculated by dividing the number of participants who complete all instruments at both time points by the total number enrolled. The intervention will be considered feasible if at least 70% of participants complete all required questionnaires.
Retention Rate (Number of Participants Remaining at 3-Month Follow-up) | Baseline and 3 months
  This outcome will measure the proportion of participants who remain enrolled in the study through the 3-month follow-up assessment. Retention will be calculated as the number of participants who complete the 3-month assessment divided by the number enrolled at baseline. Retention will be considered acceptable if at least 75% of participants remain in the study at the 3-month follow-up.
Intervention Adherence (Number of Participants Completing the Full One-Day Workshop) | 1 day
  This outcome will assess adherence to the one-day online CBT-based workshop among participants in the intervention group. The workshop consists of four modules delivered across a single day. Adherence will be defined as attending at least three of the four workshop modules. Adherence will be calculated as the number of participants meeting this criterion divided by the total number assigned to the intervention arm. The intervention will be considered feasible if at least 75% of participants meet the adherence threshold.

SECONDARY OUTCOMES:
Acceptability - TÜRBAD Satisfaction Questionnaire (TÜRBAD-SQ) | Immediately post-workshop and at 3-month follow-up
  The 6-item TÜRBAD-SQ assesses participants' satisfaction with the one-day online workshop and the perceived feasibility of the intervention procedures. The first five items use "yes/no" response options to evaluate satisfaction and feasibility, while the sixth item is open-ended and allows participants to provide additional comments. Higher proportions of "yes" responses on the closed-ended items indicate greater acceptability. The intervention will be considered acceptable if at least 70% of participants endorse "yes" on the satisfaction-related items.
Cognitive and Behavioral Change - Frequency of Actions and Thoughts Scale (FATS) | Baseline and 3 months
  The FATS is a 12-item self-report scale that measures the frequency of adaptive cognitive and behavioral skills commonly taught in Cognitive Behavioral Therapy (CBT), such as cognitive restructuring, behavioral activation, and problem solving. Items are rated on a Likert-type scale, and total scores reflect how often participants use these adaptive CBT-related thoughts and behaviors. Higher scores indicate greater use of CBT-based coping skills.
Preliminary Treatment Effect - Edinburgh Postnatal Depression Scale (EPDS) | Baseline and 3 months
  Change in EPDS scores to estimate the preliminary effect on depressive symptoms. The EPDS is a 10-item self-report measure (0-30 total score); ≥13 indicates clinically significant symptoms, and a reduction >4 points is considered clinically meaningful.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Kalaça, MD, Principal Investigator — Marmara University, Department of Psychiatry; Ayşe Sakallı Kani, MD, Study Director — Marmara University, Department of Psychiatry
Locations (1):
- Marmara University, Department of Psychiatry, Istanbul, Marmara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional and ethical restrictions. Aggregate (summary) results will be made available in related publications and presentations.

REFERENCES:
- [Background] Van Lieshout RJ, Layton H, Savoy CD, Brown JSL, Ferro MA, Streiner DL, Bieling PJ, Feller A, Hanna S. Effect of Online 1-Day Cognitive Behavioral Therapy-Based Workshops Plus Usual Care vs Usual Care Alone for Postpartum Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2021 Nov 1;78(11):1200-1207. doi: 10.1001/jamapsychiatry.2021.2488. PMID 34495285